CLINICAL TRIAL: NCT04996329
Title: A Comprehensive Tobacco Control With Early Health Warning Intervention in High Risk Population of COPD
Brief Title: Early Health Warning Intervention in Tobacco Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); Henan Provincial People's Hospital (Other); Second Hospital of Jilin University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Shandong Provincial Hospital (Other Government); Shanxi Bethune Hospital (Other); Tianjin Medical University General Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017YFC2019-255
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-04

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; brief smoking cessation intervention; current smokers; rapid decline in lung function
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- comprehensive smoking cessation intervention group (Experimental): Early health warning intervention combined with brief smoking cessation intervention Early health warning intervention is to tell the subjects that smoking leads to the rapid decline of their lung function, and they are at the high risk of developing COPD
  Interventions: Other: early health warning intervention
- brief smoking cessation intervention group (Active Comparator): brief smoking cessation intervention only
  Interventions: Other: early health warning intervention

INTERVENTIONS:
Other: early health warning intervention — early health warning intervention is to tell the subjects that smoking leads to the rapid decline of their lung function, and they are at the high risk of developing COPD.

SUMMARY:
This is a multi-center, randomized, controlled intervention clinical trial. A total of 1000 current smokers with rapid decline in lung function will be recruited and equally divided into two groups, comprehensive smoking cessation intervention group (early health warning intervention combined with brief smoking cessation intervention) and brief smoking cessation intervention group. It is aimed to evaluate whether early health warning intervention will increase the rate of smoking cessation.

DETAILED DESCRIPTION:
This is a multi-center, randomized, controlled intervention clinical trial. A total of 1,000 current smokers ( ≥ 10 pack-years) with rapid decline in lung function will be recruited from Predictive Value of Inflammatory Biomarkers and FEV1 for COPD (PIFCOPD) study (clinical trails. gov ID NCT03532893) after 1 year of follow-up. Subjects will be qually divided into two groups, comprehensive smoking cessation intervention group (early health warning intervention combined with brief smoking cessation intervention) and brief smoking cessation intervention group. Health warning intervention is to tell the subjects that smoking leads to the rapid decline of their lung function, and they are at the high risk of developing COPD. The Department of Respiratory and Critical Care of Peking University First Hospital is responsible for this research. Other 9 units participating in the study, include the The Second Hospital of Hebei Medical University, Henan Provincial People's Hospital, The Second Hospital of Jilin University, The First Affiliated Hospital of Xi'an Jiaotong University, Shandong Provincial Hospital Affiliated to Shandong University, Shan xi Dayi Hospital（Shanxi Academy of Medical Sciences）, Tianjin Medical University General Hospital, The Affiliated Hospital of Inner Mongolia University. Some questionnaire about tobacco dependence, depression, anxiety, the willingness to quit smoking and withdrawal symptoms will be collected. Exhaled CO will be measured. Subjects will recived 6 times of smoking cessation intervention in 6 month and followed in another 6 month. The primary outcome is the rate of quitting smoking. The study protocol has been approved by the Peking University First Hospital Institutional Review Board (IRB) (2019-255). Any protocol modifications will be submitted for the IRB review and approval.

ELIGIBILITY:
Inclusion Criteria:

1. aged at 40-75 years old;
2. FEV1/FVC>70% after inhaled bronchodilator
3. current smoker (≥ 10 pack-years)
4. rate of FEV1 decline >30ml/y
5. lived in a community for more than 1 years and has no plans to move out in the next 4 years

Exclusion Criteria:

1. history of asthma, COPD, lung cancer, active pulmonary tuberculosis, bronchiectasis, diffuse lung disease (interstitial pneumonia, pulmonary sarcoidosis, occupational lung disease, sarcoidosis et al) and pleural disease;
2. history of lobectomy and / or lung transplantation;
3. predicted life expectancy less than 3 years;
4. history of severe psychiatric illnesses, mental disorders, neurological disorders, malignant tumors, chronic liver disease, heart failure, autoimmune diseases, chronic kidney disease;
5. Alcoholism, drug abuse or abuse of toxic solvents;
6. Cannot finish long term follow-up or poor compliance;
7. Do not provide consent

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of quitting smoking | 1 year
  keep smoking cessation for more than 6 months

SECONDARY OUTCOMES:
one month smoking cessation rate | 6 months
  stop smoking for more than one month, but less than six months
smoking reduction rate | 1 year
  less than the number of cigarettes before the first intervention
smoking cessation rate at each follow-up | 6 months
  stop smoking for 24 hours or more
relapse rate | 1 year
  relapse rate of smoking

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The Second Hospital of Jilin University, Ch’ang-ch’un
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - Shandong Provincial Hospital Affiliated to Shandong University, Jing’an
  - The First Hospital of Qinhuangdao, Qinhuangdao
  - The Second Hospital of Hebei Medical University, Shijia Zhuang
  - Shanxi Bethune Hospital, Taiyuan
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Henan Provincial People's Hospita, Zhenzhou

IPD SHARING:
Plan to Share IPD: No